CLINICAL TRIAL: NCT02518139
Title: A Phase 3, 52-week, Randomized, Active-Controlled Parallel Group Study to Evaluate the Safety and Tolerability of Nebulized TD-4208 in Subjects With Chronic Obstructive Pulmonary Disease
Brief Title: A 52-Week Parallel Group Safety Study of TD-4208 in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mylan Inc. (Industry)
Collaborators: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0128
Record Dates: First submitted 2015-08-05; First posted 2015-08-07 (Estimated); Results first posted 2018-12-31 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Chronic Obstructive Pulmonary Disease, COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — revefenacin; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- TD-4208-1 (Experimental): 88 mcg
  Interventions: Drug: TD-4208
- TD-4208-2 (Experimental): 175 mcg
  Interventions: Drug: TD-4208
- Tiotropium (Active Comparator): 18 mcg
  Interventions: Drug: Tiotropium

INTERVENTIONS:
Drug: TD-4208 — Subjects receiving TD-4208 are blinded to one of two doses of 4208.
  Other Names: revefenacin
  Arms: TD-4208-1; TD-4208-2
Drug: Tiotropium — There is not a placebo, there is an active comparator (Tiotropium) arm.
  Arms: Tiotropium

SUMMARY:
The purpose of this study is to measure the safety and tolerability of TD 4208, an investigational drug being developed to treat people with moderate to very severe COPD, compared to tiotropium.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a male or female subject 40 years of age or older

Exclusion Criteria:

* Females who are pregnant, lactating, breast-feeding or planning to become pregnant during the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1060 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma
Locations (1):
- Palmetto Medical Research Associates L.L.C, Easley, South Carolina, United States

REFERENCES:
- [Derived] Ohar JA, Mahler DA, Davis GN, Lombardi DA, Moran EJ, Crater GD. Clinical Burden of Chronic Obstructive Pulmonary Disease in Patients with Suboptimal Peak Inspiratory Flow. Can Respir J. 2024 Mar 22;2024:8034923. doi: 10.1155/2024/8034923. eCollection 2024. PMID 38560416
- [Derived] Barnes CN, Mahler DA, Ohar JA, Lombardi DA, Crater GD. Peak Inspiratory Flows: Defining Repeatability Limits and a Predictive Equation for Different Inhalers. Chest. 2020 Oct;158(4):1413-1419. doi: 10.1016/j.chest.2020.03.072. Epub 2020 Apr 25. PMID 32343967
- [Derived] Donohue JF, Kerwin E, Sethi S, Haumann B, Pendyala S, Dean L, Barnes CN, Moran EJ, Crater G. Maintained therapeutic effect of revefenacin over 52 weeks in moderate to very severe Chronic Obstructive Pulmonary Disease (COPD). Respir Res. 2019 Oct 30;20(1):241. doi: 10.1186/s12931-019-1187-7. PMID 31666076
- [Derived] Donohue JF, Kerwin E, Sethi S, Haumann B, Pendyala S, Dean L, Barnes CN, Moran EJ, Crater G. Revefenacin, a once-daily, lung-selective, long-acting muscarinic antagonist for nebulized therapy: Safety and tolerability results of a 52-week phase 3 trial in moderate to very severe chronic obstructive pulmonary disease. Respir Med. 2019 Jul;153:38-43. doi: 10.1016/j.rmed.2019.05.010. Epub 2019 May 23. PMID 31150963

RESULTS

PARTICIPANT FLOW:
Groups:
- TD-4208-1: 88 mcg
  TD-4208: There is not a placebo, there is a comparator (Tiotropium) arm, and the subjects are blinded to one of two doses of 4208 or un-blinded to Tiotropium.
- TD-4208-2: 175 mcg
  TD-4208: There is not a placebo, there is a comparator (Tiotropium) arm, and the subjects are blinded to one of two doses of 4208 or un-blinded to Tiotropium.
- Tiotropium: 18 mcg
  Tiotropium: Active comparator
Period: Overall Study
Arm/Group | TD-4208-1 | TD-4208-2 | Tiotropium
Started | 364 | 335 | 356
Completed | 219 | 191 | 262
Not Completed | 145 | 144 | 94

BASELINE CHARACTERISTICS:
Population: 1060 subjects were randomized. A total of 1055 subjects received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | TD-4208-1 | TD-4208-2 | Tiotropium | Total
Number analyzed (Participants) | 364 | 335 | 356 | 1055
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 183 | 167 | 163 | 513
  >=65 years | 181 | 168 | 193 | 542
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (9.36) | 64.4 (8.61) | 64.9 (8.91) | 64.4 (8.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 158 | 139 | 142 | 439
  Male | 206 | 196 | 214 | 616
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 5 | 3 | 14
  Not Hispanic or Latino | 357 | 326 | 352 | 1035
  Unknown or Not Reported | 1 | 4 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 24 | 21 | 24 | 69
  White | 337 | 309 | 331 | 977
  More than one race | 1 | 2 | 0 | 3
  Unknown or Not Reported | 1 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 364 | 335 | 356 | 1055
Smoking Status [Count of Participants; unit: Participants]
  Current Smoker | 171 | 151 | 167 | 489
  Former Smoker | 193 | 184 | 189 | 566

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events: Frequency and Severity
Description: To assess the safety and tolerability of TD-4208 by assessing the frequency and severity of Treatment Emergent Adverse Events (TEAE)
Time Frame: Baseline to Day 365
Measure: Count of Participants; unit: Participants
Groups:
- TD-4208-1: 88 mcg
  TD-4208
- TD-4208-2: 175 mcg
  TD-4208
Arm/Group | TD-4208-1 | TD-4208-2 | Tiotropium
Number analyzed (Participants) | 364 | 335 | 356
Participants
  Adverse Event (AE) | 272 | 242 | 275
  Moderate or Severe AE | 226 | 174 | 210
  Serious AE | 58 | 43 | 58

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from signing of the ICF through the final follow-up assessment (approximately 1 year)
Arm/Group | TD-4208-1 | TD-4208-2 | Tiotropium
All-Cause Mortality (participants affected / at risk) | 1/364 | 1/335 | 1/356
Serious Adverse Events (participants affected / at risk) | 58/364 | 43/335 | 58/356
Other Adverse Events (participants affected / at risk) | 202/364 | 166/335 | 188/356
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TD-4208-1 (N=364) | TD-4208-2 (N=335) | Tiotropium (N=356)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 8 (8) | 13 (13)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 10 (10) | 1 (1) | 6 (6)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 2 (2)
Lung adenocarcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 3 (3) | 2 (2)
Myocardial infarction (Cardiac disorders) | 4 (4) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0) | 3 (3)
Angina unstable (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal angiodysplasia haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatic mass (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 3 (3) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
Impaired healing (General disorders) | 0 (0) | 1 (1) | 1 (1)
Cardiac death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Device malfunction (General disorders) | 0 | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Near drowning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Nerve compression (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Accelerated hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertensive emergency (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Bipolar I disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Abscess neck (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis intestinal haemorrhagic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Fungaemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infected skin ulcer (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Ludwig angina (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Peritoneal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Colon cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Ear neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Laryngeal squamouse cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lung adenocarcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Small initestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TD-4208-1 (N=364) | TD-4208-2 (N=335) | Tiotropium (N=356)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 107 (107) | 73 (73) | 100 (100)
Nasopharyngitis (Infections and infestations) | 28 (28) | 26 (26) | 17 (17)
Upper Respiratory Tract Infection (Infections and infestations) | 24 (24) | 20 (20) | 24 (24)
Cough (Respiratory, thoracic and mediastinal disorders) | 18 (18) | 25 (25) | 20 (20)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 31 (31) | 13 (13) | 13 (13)
Headache (Nervous system disorders) | 15 (15) | 13 (13) | 20 (20)
Urinary tract infection (Infections and infestations) | 20 (20) | 11 (11) | 15 (15)
Bronchitis (Infections and infestations) | 17 (17) | 17 (17) | 9 (9)
Hypertension (Vascular disorders) | 18 (18) | 8 (8) | 16 (16)
Diarrhoea (Gastrointestinal disorders) | 14 (14) | 13 (13) | 9 (9)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 16 (16) | 5 (5) | 14 (14)
Sinusitis (Infections and infestations) | 15 (15) | 8 (8) | 9 (9)
Back Pain (Musculoskeletal and connective tissue disorders) | 10 (10) | 7 (7) | 10 (10)
Anthralgia (Musculoskeletal and connective tissue disorders) | 9 (9) | 6 (6) | 11 (11)
Nausea (Gastrointestinal disorders) | 7 (7) | 6 (6) | 12 (12)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 8 (8) | 8 (8) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI may communicate the trial results generated by the PI, but only after the first publication or presentation of the combined study results generated by all participating sites. The Sponsor can then review trial results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days. The Sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2016-01-21): https://cdn.clinicaltrials.gov/large-docs/39/NCT02518139/Prot_001.pdf
  • Statistical Analysis Plan (2017-03-13): https://cdn.clinicaltrials.gov/large-docs/39/NCT02518139/SAP_000.pdf